CLINICAL TRIAL: NCT07229495
Title: Efficacy and Safety of Tegileridine for Postoperative Analgesia Following Adolescent Scoliosis Correction Surgery: A Prospective, Single-Center, Double-Blind, Non-Inferiority, Randomized Controlled Trial
Brief Title: Tegileridine for Postoperative Pain After Adolescent Scoliosis Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lan Ling, Principal Investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K7767
Record Dates: First submitted 2025-09-24; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis; Adolescence; Pain After Surgery; Analgesia, Patient-controlled
Keywords: Tegileridine; Postoperative Pain; Adolescent; Patient-Controlled Analgesia; Scoliosis
MeSH Terms: conditions — Scoliosis; Agnosia; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegileridine 1 μg/kg PCA (Experimental): Participants in this arm will receive Tegileridine for postoperative patient-controlled analgesia (PCA). The intervention is administered as an intravenous infusion via a PCA pump. The PCA solution is prepared by diluting Tegileridine injection in normal saline to a total volume of 100 ml. The bolus dose is 1 μg/kg of Tegileridine per activation, with no background infusion. The lockout interval between bolus doses is 10 minutes. PCA therapy will be initiated in the post-anesthesia care unit (PACU) immediately after surgery and maintained for at least 48 hours, barring any PCA-related adverse events requiring discontinuation.
  Interventions: Drug: Tegileridine
- Tegileridine 2 μg/kg PCA (Experimental): Participants in this arm will receive Tegileridine for postoperative patient-controlled analgesia (PCA). The intervention is administered as an intravenous infusion via a PCA pump. The PCA solution is prepared by diluting Tegileridine injection in normal saline to a total volume of 100 ml. The bolus dose is 2 μg/kg of Tegileridine per activation, with no background infusion. The lockout interval between bolus doses is 10 minutes. PCA therapy will be initiated in the post-anesthesia care unit (PACU) immediately after surgery and maintained for at least 48 hours, barring any PCA-related adverse events requiring discontinuation.
  Interventions: Drug: Tegileridine
- Morphine 20 μg/kg PCA (Active Comparator): Participants in this arm will receive Morphine for postoperative patient-controlled analgesia (PCA). This arm serves as the active comparator. The intervention is administered as an intravenous infusion via a PCA pump. The PCA solution is prepared by diluting Morphine injection in normal saline to a total volume of 100 ml. The bolus dose is 20 μg/kg of Morphine per activation, with no background infusion. The lockout interval between bolus doses is 10 minutes. PCA therapy will be initiated in the post-anesthesia care unit (PACU) immediately after surgery and maintained for at least 48 hours, barring any PCA-related adverse events requiring discontinuation.
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: Tegileridine — Tegileridine is an investigational novel opioid receptor agonist. In this study, it is administered as an intravenous infusion via a patient-controlled analgesia (PCA) pump for postoperative pain management. The PCA solution is prepared by diluting Tegileridine injection in normal saline.
  Arms: Tegileridine 1 μg/kg PCA; Tegileridine 2 μg/kg PCA
Drug: morphine — Morphine is a standard opioid analgesic used as the active comparator in this study. It is administered as an intravenous infusion via a patient-controlled analgesia (PCA) pump for postoperative pain management. The PCA solution is prepared by diluting Morphine injection in normal saline.
  Arms: Morphine 20 μg/kg PCA

SUMMARY:
The goal of this clinical trial is to see if a new pain medicine called Tegileridine is at least as effective as morphine (the standard treatment) for pain relief after spinal surgery in teenagers with scoliosis. This type of study is called a "non-inferiority" trial. The study will also carefully compare the safety of both medicines.

The main questions it aims to answer are:

Is Tegileridine no worse than morphine at controlling pain in the first 24 hours after surgery? How do the side effects (like sleepiness or nausea) of Tegileridine compare to those of morphine? Researchers will compare two different doses of Tegileridine against morphine. Neither the participants nor the doctors assessing them will know which medicine is being given.

Participants in this study will:

Receive one of the three pain medicine options through a pump (called a PCA pump) that they can control themselves after surgery.

Use the pump for up to 48 hours. Regularly rate their pain levels using a simple number scale. Have their health closely monitored by the study team during this time.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double-blind, controlled, non-inferiority clinical trial designed to evaluate the efficacy and safety of Tegileridine for postoperative patient-controlled analgesia (PCA) in adolescent patients undergoing spinal fusion surgery for scoliosis.

Postoperative pain management is crucial for recovery, with opioids like morphine being the standard of care. However, morphine is associated with significant side effects, including respiratory depression, nausea, and vomiting. Tegileridine is a novel, highly selective μ-opioid receptor agonist that is hypothesized to provide potent analgesia with an improved safety profile, particularly regarding respiratory depression.

A total of 171 adolescent patients (aged 10 to <18 years) scheduled for surgery will be enrolled. Participants will be randomly assigned in a 1:1:1 ratio to one of three treatment groups:

Group T1: Tegileridine PCA at a dose of 1 μg/kg per bolus. Group T2: Tegileridine PCA at a dose of 2 μg/kg per bolus. Group M (Active Comparator): Morphine PCA at a dose of 20 μg/kg per bolus. The study medication will be prepared by an unblinded nurse not involved in subsequent patient care or assessment. The PCA pump will be initiated upon arrival in the post-anesthesia care unit (PACU) after surgery and will be maintained for 48 hours. To maintain blinding, the study drugs are diluted in normal saline to appear identical. Patients, attending anesthesiologists, and outcome assessors will all be blinded to the treatment assignment.

The primary objective is to demonstrate the non-inferiority of Tegileridine to morphine in terms of analgesic efficacy. The primary efficacy endpoint is the area under the curve (AUC) of resting pain intensity scores, measured on an 11-point Numerical Rating Scale (NRS), over the first 24 hours after initiating PCA. A predefined non-inferiority margin of 12 will be used for the comparison. Statistical testing will follow a hierarchical procedure, first comparing the T2 group to the morphine group, and if non-inferiority is established, proceeding to compare the T1 group to morphine.

Secondary objectives include comparing the groups on various efficacy measures, such as pain AUC at other time points, rescue analgesic consumption, and patient satisfaction. Safety objectives focus on the incidence and severity of adverse events, with continuous monitoring for postoperative hypoxemia (SpO₂ < 90%), assessment of sedation levels using the modified Pasero Opioid-induced Sedation Scale (m-POSS), and recording of other common opioid-related side effects like postoperative nausea and vomiting (PONV).

The primary analysis will be conducted on the Full Analysis Set (FAS). Sensitivity analyses and a pre-specified subgroup analysis by gender are also planned.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 years to less than 18 years.
* Scheduled to undergo posterior spinal fusion (PSF) surgery for scoliosis under general anesthesia.
* American Society of Anesthesiologists (ASA) physical status classification I to III.
* The participant and their parent or legal guardian voluntarily provide written informed consent prior to any study-related procedures.

Exclusion Criteria:

* History of difficult airway, severe respiratory depression (SpO₂ < 90%), acute or severe bronchial asthma.
* History of severe cardiovascular or cerebrovascular disease, such as myocardial infarction, unstable angina, second-degree or higher atrioventricular block, NYHA Class III or higher heart failure, or stroke.
* Known or suspected gastrointestinal obstruction, including paralytic ileus.
* Known hypersensitivity to opioids or any component of the study drug formulation.
* History of psychiatric disorders (e.g., schizophrenia, depression) or cognitive impairment.
* Diagnosis of neuromuscular scoliosis or presence of any other chronic pain condition that may interfere with postoperative pain assessment.
* Chronic use of opioid analgesics or use of any analgesic medication within 48 hours prior to surgery.
* Planned postoperative admission to the intensive care unit (ICU).
* Any other condition deemed by the investigator to be inappropriate for participation in the study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of Resting Pain Scores on the 11-point Numerical Rating Scale (NRS) Over the First 24 Hours Postoperative | From the initiation of Patient-Controlled Analgesia (PCA) up to 24 hours post-initiation.
  The analgesic efficacy will be assessed by calculating the Area Under the Curve (AUC) of the resting pain intensity scores over the first 24 hours after initiating Patient-Controlled Analgesia (PCA).
  Pain Intensity Measurement: Pain intensity is assessed by the participant using an 11-point Numerical Rating Scale (NRS), where 0 represents "no pain" and 10 represents "the worst pain imaginable." Resting state is defined as being in a stationary position without active movement.
  Assessment Time Points: NRS scores are recorded at predefined time points: 5 minutes, 10 minutes, 15 minutes, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, and 24 hours after PCA initiation.
  AUC Calculation: The AUC for the NRS scores versus time is calculated using the trapezoidal rule, which sums the areas of trapezoids formed between consecutive time points. A lower AUC indicates better and more sustained pain control over the 24-hour period.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of Resting Pain Scores on the Numerical Rating Scale (NRS) Over Multiple Time Intervals | The AUC will be calculated for the cumulative intervals from PCA initiation up to 6 hours, 12 hours, and 48 hours post-initiation.
  The AUC of resting pain intensity scores (measured on an 11-point NRS, where 0 represents "no pain" and 10 represents "the worst pain imaginable") will be calculated using the trapezoidal rule. The AUC will be calculated for the following cumulative time intervals after PCA initiation: 0-6 hours, 0-12 hours, and 0-48 hours. A lower AUC indicates better and more sustained pain control over the specified period.
Area Under the Curve (AUC) of Activity-Induced Pain Scores on the Numerical Rating Scale (NRS) over Multiple Intervals | Assessed at 6, 12, 24, and 48 hours after PCA initiation.
  The AUC of pain intensity scores during activity (or coughing) measured on an 11-point NRS will be calculated over the intervals of 0-6 hours, 0-12 hours, 0-24 hours, and 0-48 hours after PCA initiation. The AUC is calculated using the trapezoidal rule.
Resting and Activity-Induced Pain Scores on the Numerical Rating Scale (NRS) at Multiple Time Points | Assessed at 16 predefined time points from 5 minutes to 48 hours after PCA initiation.
  Pain intensity will be assessed using the 11-point NRS (0=no pain, 10=worst pain imaginable) at rest and during activity (or coughing) at the following time points after PCA initiation: 5 minutes, 10 minutes, 15 minutes, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 30 hours, 36 hours, 42 hours, and 48 hours.
Proportion of Participants Requiring Rescue Analgesia | From PCA initiation up to 48 hours post-initiation.
  The percentage of participants who receive rescue analgesia during the PCA treatment period. Rescue analgesia is defined as the administration of additional analgesic medication (e.g., acetaminophen, NSAIDs, or other opioids) when the participant's pain is not adequately controlled (NRS score ≥4) despite receiving the study drug.
Time to First Use of Rescue Analgesia | From PCA initiation up to 48 hours post-initiation (time to event is measured).
  The time elapsed from the initiation of the PCA pump to the first administration of any rescue analgesic medication.
Total Number of Rescue Analgesic Administrations Per Participant | From PCA initiation up to 48 hours post-initiation.
  The total count of rescue analgesic medication administrations required for each participant during the PCA treatment period, when pain was not controlled (NRS ≥4) by the study drug.
Cumulative Dose of Rescue Analgesic Medication | From PCA initiation up to 48 hours post-initiation.
  The total cumulative dose of all rescue analgesic medications used by each participant during the PCA treatment period. Doses of different opioids will be converted to morphine milligram equivalents (MME) for summation.
Proportion of Participants with Pain NRS Score ≤ 3 at Each Assessment Time Point | Assessed at 16 predefined time points from 5 minutes to 48 hours after PCA initiation.
  The percentage of participants who achieve a pain intensity score of 3 or less (indicating mild pain) on the 11-point NRS at the following time points after PCA initiation: 5 minutes, 10 minutes, 15 minutes, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 18 hours, 24 hours, 30 hours, 36 hours, 42 hours, and 48 hours.
Total Number of PCA Pump Attempts and Successful Deliveries | From PCA initiation up to 48 hours post-initiation.
  The total number of demands (attempts) made by the participant on the PCA pump and the total number of successful drug deliveries (effective deliveries) recorded by the pump during the treatment period.
Postoperative Length of Hospital Stay | From the day of surgery to the day of hospital discharge, an average of 10 days.
  The duration of hospitalization after the surgical procedure, measured from the day of surgery until the day of discharge.
Satisfaction with Pain Treatment | At 30 minutes after stopping PCA (typically around 48 hours post-surgery).
  Participants' satisfaction with pain management is assessed using an 11-point numerical scale (0=extremely dissatisfied, 10=extremely satisfied) within 30 minutes after the cessation of PCA therapy.
Incidence of Postoperative Hypoxemia | From PCA initiation up to 48 hours post-initiation.
  The proportion of participants experiencing postoperative hypoxemia, defined as a percutaneous oxygen saturation (SpO2) reading below 90%, as monitored by pulse oximetry during the PCA treatment period.
Incidence and Severity of Postoperative Nausea and Vomiting (PONV) | Assessed at 5 minutes, 10 minutes, 30 minutes, 6 hours, 12 hours, 18 hours, 24 hours, 36 hours, and 48 hours after PCA initiation.
  The occurrence and severity of PONV assessed by healthcare personnel using a Visual Analog Scale (VAS) for nausea/vomiting (0=no nausea/vomiting, 10=worst imaginable nausea/vomiting) at specified time points. Severity is categorized as mild (VAS<4cm), moderate (VAS 4-7cm), or severe (VAS>7cm).
Level of Sedation as Assessed by the Modified Pasero Opioid-Induced Sedation Scale (m-POSS) | Assessed at 5 minutes, 10 minutes, 30 minutes, 6 hours, 12 hours, 18 hours, 24 hours, 36 hours, and 48 hours after PCA initiation.
  The level of sedation is assessed by healthcare personnel using the m-POSS, which includes scores from S (sleep, easily aroused) to 4 (somnolent, minimal or no response to stimulus). Higher scores indicate deeper sedation.
Incidence of Other Adverse Events | From PCA initiation up to 48 hours post-initiation.
  The occurrence of other predefined adverse events during the treatment period, including abdominal pain, abdominal distension (time to first flatus and defecation), fever, dizziness, headache, sinus bradycardia, somnolence, and pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Lan, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share Individual Participant Data (IPD) from this trial. The primary reason is to ensure the confidentiality of the participants, who are adolescents. Any future consideration of data sharing would require approval from the relevant ethics committee and would only proceed after the data has been de-identified to a standard that fully protects participant privacy.